CLINICAL TRIAL: NCT03074812
Title: Exploring Mechanisms for Neuropsychiatric Symptoms of Parkinson Disease Using Transcranial Direct Current Stimulation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding and did not complete enrollment.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00087957
Record Dates: First submitted 2016-03-02; First posted 2017-03-09 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Idiopathic Parkinson's Disease; Parkinson Disease; Depression
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — Transcranial Direct Current Stimulation; Deep Brain Stimulation; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham tDCS (Sham Comparator): Sham transcranial direct current stimulation where current will be reduced to zero after standardized ramp up to 2 mA
  Interventions: Device: Transcranial Direct Current Stimulation
- Active tDCS (Experimental): Transcranial direct current stimulation according to protocol maintained for 30 minutes after ramping up to 2 mA
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial direct current stimulation (tDCS) is a commonly used non-invasive form of brain stimulation for studying motor functions in health and disease [36]. It involves the attachment of surface electrodes to the scalp through which very small electric currents (1 or 2mA) are applied via a current regulated device. The currents do not produce any sensation. The applied current affects excitability of underlying neural tissue.
  Other Names: tDCS; Brain Stimulation; Neuromodulation

SUMMARY:
This study evaluates the effect of transcranial direct current stimulation (tDCS) on non-motor symptoms of Parkinson's disease, including depression and cognitive symptoms. Participants are randomized to receive active or sham tDCS for 30 minutes over 10 treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* Abel to provide written informed consent is obtained in the English language
* Age 18 to 95 years old
* Movement Disorder Society Clinical Diagnostic Criteria for probable idiopathic Parkinson disease
* Report disabling depressive or neuropsychiatric symptoms prior to study entry
* Capacity to understand the nature of the study;

Exclusion Criteria:

* Known structural brain disease such as a neoplasm, abscess etc.
* Pre-existing skull / scalp defects that would impede standardized electrode placement
* Current electronic or metal implants
* Diagnosis of Bipolar Disorder, Post-Traumatic Stress Disorder, a Psychotic Disorder or any other non-unipolar depressive disorder as a principal diagnosis in the 6 months prior to screening;
* Concurrent treatment with medication which may affect tDCS (benzodiazepines, anticonvulsants, dextromethorphan and pseudoephedrine)
* Endorse active suicidal ideation at enrollment or during any study visit, or have attempted suicide in the six months prior to screening;
* History of substance abuse or dependence in the 2 months prior to screening;
* Considered to be at significant risk of committing homicide;
* Unstable medical condition;
* Score less than 22 on the Montreal Cognitive Assessment (MoCA)
* Women of childbearing potential who are pregnant or are considering becoming pregnant during the length of the study;
* There has been a change in their depression or psychotherapy treatment regimen in the 2 weeks preceding screening;

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Demonstrating improvements on Objective Rating Scales of Depression via structured interview | 1 months
  Primary outcome measure will be the number of participants who demonstrate remission of depressive symptoms OR improvement of 50% (i.e. response) on the Montgomery-Asberg Scale of Depression (MADRS)

SECONDARY OUTCOMES:
Apathy Scores as measure by a self-report scale (the Apathy Scale) | 1 months
  The dimensional degree of change in Apathy symptoms as assessed via the Apathy Scale, a subjective self-report tool of apathetic symptoms
Subjective Depression Severity rated via self-report on depression inventory | 1 months
  Subjective severity of depression as measured via self-reported Beck Depression Inventory - II
Subjective reactive to pleasure (i.e. improvement of anhedonia) as rated via self-report | 1 month
  Monitoring degree of change of hedonic-tone scores via the Snaith-Hamilton Pleasure Scale (SHAPS)
Subjective improvement of Anxiety Symptoms via Rating Scale | 1 month
  The change in Parkinson Anxiety Scale (PAS) score per person and across sham v. experimental groups.
Performance on abbreviated cognitive battery | 1 month
  Objective improvement on measures of attention, verbal fluency, working memory and recall by various bedside cognitive tests
Improvement of Parkinsonian Motor Symptoms | 1 month
  Number of participants between arms and individual improvement of Movement Disorders Society Unified Parkinson Disease Rating Scale Part 3 (MDS-UPDRS Pt3) Score.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Mills, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital / Johns Hopkins University, Baltimore, Maryland, United States